CLINICAL TRIAL: NCT04412967
Title: A Randomized, Controlled Comparison of Nurse-led Placement of Peripheral Venous Catheters in Overweight Patients Using Standard or Dynamic Ultrasound-guided Technique
Brief Title: Nurse-led Placement of Peripheral Venous Catheters in Overweight Patients Using Standard or Dynamic Ultrasound-guided Technique
Acronym: DUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, Principal Investigator, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SE-2020 JG DUST
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Overweight and Obesity; Emergencies
Keywords: Nurse led; Ultrasound; Emergency department; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Technique PVC placement (Active Comparator): Standard PVC placement technique
  Interventions: Other: Standard technique of placing a PVC
- DUST (Experimental): Dynamic ultrasound-guided short-axis needle tip navigation (DUST)
  Interventions: Device: Dynamic ultrasound-guided short-axis needle tip navigation

INTERVENTIONS:
Device: Dynamic ultrasound-guided short-axis needle tip navigation — placement of peripheral venous catheters using ultrasound guided technique
  Arms: DUST
Other: Standard technique of placing a PVC — Standard technique with palpation or Visual inspection of the pvc placement site
  Arms: Standard Technique PVC placement

SUMMARY:
Overweight and obesity may be associated with difficult intravenous access leading to longer procedure time and more placement attempts of peripheral venous catheters (PVC). Dynamic ultrasound-guided short-axis needle tip navigation (DUST) may facilitate the procedure.

This was a prospective, randomized, non-blinded study to compare time and placement attempts for nurse-led standard (ST) and ultrasound guided PVC placement in 90 emergency patients with a BMI ≥25kg/m2.

Consenting patients were randomized at a 1:1 ratio to receive PVC by either ST or DUST.

Application time was defined as the time from applying stasis to visible blood in the PVC flash-chamber.

No difference in time was found (medians: ST 42 s; DUST 53.5 s, P = 0.535). There were on average 17 % less placement attempts in the DUST-group (median 1 attempt; Q1 = 1 Q3 = 1) compared to the ST-group (median 1 attempt; Q1 = 1 Q3 = 1.5), (p = 0.031). Patients reported no differences in perceived pain (p = 0.955) or perceived satisfaction (p = 0.342). Pain and subcutaneous infiltrations were the only side-effects reported (ST-group 6, DUST-group 5).

DUST does not decrease time to functional PVC but reduces the number of PVC placement attempts in patients with BMI ≥25 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* REETS prioritization level of "Orange", "Yellow", "Green" or "Blue"
* 18 years old
* BMI ≥25 Kg/m2
* Need of PVC according to Emergency department guidelines
* Able to give written informed consent

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Life threatening patient status (REETS prioritization level of "Red")
* Immunosuppression
* Pregnant or lactating women
* Blood infections
* Puncture zone skin damaged (burns, eczema, infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-06-03 (Actual)

PRIMARY OUTCOMES:
Time to application | 1 hour
  Application time was defined as the time from applying stasis to visible blood in the PVC flash-chamber.
Number of cannulation attempts | 1 hour
  The total number of cannulation attempts performed per patient

SECONDARY OUTCOMES:
Patient satisfaction | 1 hour
  The perceived satisfaction of the patient as indicated by Numeric Rating scale (NRS, 0 = not satisfied, 10 = maximum satisfaction)
Perceived Pain | 1 hour
  The perceived pain of the patient as indicated by Numeric Rating scale (NRS, 0 = no pain, 10 = the worst pain possible)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wilhelms, Phd, Principal Investigator — Linkoeping University
Locations (1):
- University Hospital Linköping, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04412967/ICF_000.pdf